CLINICAL TRIAL: NCT03632616
Title: Quality of Life Evaluation of Endoscopic Interventions in Chronic Pancreatitis
Brief Title: Quality of Life Assessment of Chronic Pancreatitis Endoscopic Interventions
Acronym: QOLAPI
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1816
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; quality of life
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PANQOLI (quality of life instrument) — A quality of life instrument, the PANQOLI, will be administered prior to endoscopic intervention, and at 1,3, 6 and 12 months post-intervention.
  Other Names: Visual Analog Scale for pain

SUMMARY:
This study seeks to evaluate the effect of endoscopic interventions on quality of life in patients with chronic pancreatitis. Quality of life will be evaluated using the PANQOLI, a validated quality of life instrument specific to chronic pancreatitis. Endoscopic interventions will include pancreatic duct dilation and stenting, celiac plexus block, lithotripsy and removal of pancreatic duct stones, and pseudocyst drainage.

DETAILED DESCRIPTION:
This is a multicenter prospective cohort study assessing the impact of endoscopic interventions on patients with chronic pancreatitis. Patients with chronic pancreatitis referred for endoscopic treatment, including pancreatic duct dilation and stenting, pseudocyst drainage, celiac plexus blocks, and pseudocyst drainage/necrosectomy will be enrolled in this study. They will receive a baseline evaluation using the PANQOLI, a chronic pancreatitis-specific quality of life instrument, in addition to a visual analog scale to measure their pain. Demographic and endoscopic features will be collected in addition to pain medication use. Patients will receive follow-up at 1, 3, and 6 months post-intervention consisting of the PANQOLI, visual analog scale for pain, and pain medication use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful chronic pancreatitis, defined as either 1) the presence of pancreatic calcifications on cross-sectional imaging, 2) morphologic changes consistent with the Rosemont criteria on endoscopic ultrasound, or 3) endoscopic pancreatic function test results consistent with decreased pancreatic function.

Exclusion Criteria:

* Pregnant females
* Prisoners
* Patients under the age of 18
* Patients lacking the capacity to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with painful chronic pancreatitis who are being referred for endoscopic treatment to reduce their pain.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life using the PANQOLI (PANcreatitis Quality of Life Instrument) | The outcome will be measured at 1, 3, and 6 months post-intervention.
  The primary outcome will be the change in quality of life using the PANQOLI (PANcreatitis Quality of Life Instrument) after endoscopic intervention.

SECONDARY OUTCOMES:
Change in pain level using the Visual Analog Scale (VAS) for pain. | The outcome will be measured at 1, 3, and 6 months post-intervention.
  The secondary outcome will include the change in pain using the Visual Analog Scale (VAS) for pain after endoscopic intervention
Change in pain medication use | The outcome will be measured at 1, 3, and 6 months post-intervention.
  The secondary outcome will include the change in pain medication use after endoscopic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Raj J Shah, MD, Principal Investigator — Professor of Medicine; Director, Pancreas and Biliary Endoscopy
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Center, Aurora, Colorado
  - Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No